CLINICAL TRIAL: NCT03946098
Title: Implementation of Internet-based Cognitive Behavior Therapy for Problem Gambling in Routine Addiction Care: A Feasibility Study
Brief Title: ICBTG in Routine Care
Acronym: iCBTG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Anne H Berman, Associate professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0428
Record Dates: First submitted 2019-04-28; First posted 2019-05-10 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Problem Gambling; Gambling Disorder
Keywords: Internet intervention; Gambling Disorder; Cognitive-behavioral therapy; Psychiatric comorbidity; Regular addiction care; Problem gambling
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iCBT for Gambling Disorder (Experimental): Treatment will consist of a 1+10 module internet delivered CBT program targeting problem gambling, newly developed. A bottom-up procedure was used to develop the treatment protocol, inspired by Clark's (2004) method for developing novel CBT treatments. We developed a clinical model delineating what factors contribute to the persistence of problem gambling behavior, and aligned these with targeted treatment interventions; based on behavioral upon research on the learning and maintenance processes of gambling behavior (Ramnerö et al, in press), theoretical models of gambling and comorbidity (Blaszczynski & Nower, 2002); as well as qualitative interviews with treatment seeking gamblers with or without comorbidity.
  Interventions: Behavioral: iCBT

INTERVENTIONS:
Behavioral: iCBT — A newly developed iCBT protocol targeting problem gambling.

SUMMARY:
Problem gambling (PG) is a major public health concern worldwide. As awareness of PG has risen, treatment demand is increasing, and internet interventions is a promising alternative for providing fast, evidence-based treatment at scale, to a low cost. This article presents the protocol of an open label, uncontrolled pilot and feasibility trial of a novel internet-delivered cognitive behavioral treatment, conducted in regular addiction care with adult treatment-seeking patients (max N=25) with problematic gambling. Weekly measures of gambling symptoms and gambling will serve as outcome measures. Study results will further guide the development of the intervention and its implementation into regular addiction care.

ELIGIBILITY:
Inclusion criteria:

* being at least 18 years old
* living in Sweden
* being able to read and write Swedish.
* having a total score of >= 3 on the Problem Gambling Severity Index (PGSI; Ferris & Wynne, 2001)
* having the ability to work with online treatment material by themselves (with support from a therapist)

Exclusion criteria:

* fulfilling criteria for ongoing manic episode
* currently undergoing a parallel CBT treatment for Gambling Disorder or problem gambling.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2021-02-09 (Actual); Study Completion 2021-02-09 (Actual)

PRIMARY OUTCOMES:
The Gambling Symptom Assessment Scale (G-SAS) | Past 7 days
  Gambling symptoms

SECONDARY OUTCOMES:
The Gambling Time Line Follow Back (TLFB-G) | Past 7 days
  Gambling behavior
The 9-item Patient Health Questionnaire (PHQ-9 | Past 2 weeks
  Depressive symptoms
The 7-item Generalised Anxiety Disorder scale (GAD-7) | Past 2 weeks
  Anxiety symptoms
The Alcohol Use Disorders Identification Test (AUDIT) | Past 12 months
  Alcohol use
The Drug Use Disorders Identification Test (DUDIT) | Past 12 months
  Drug use
the 26-item World Health Organization Quality of Life-BREF (WHOQOL-BREF) | Past 2 weeks
  Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Philip H Lindner, PhD, Study Chair — Karolinska Institutet
Locations (1):
- eStöd, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Molander O, Lindner P, Ramnero J, Bjureberg J, Carlbring P, Berman AH. Internet-based cognitive behavior therapy for problem gambling in routine care: protocol for a non-randomized pilot and feasibility trial. Pilot Feasibility Stud. 2020 Jul 21;6:106. doi: 10.1186/s40814-020-00647-5. eCollection 2020. PMID 32699645